CLINICAL TRIAL: NCT02652754
Title: Open Label Pharmacokinetic Study of Granexin® Gel in Patients With Diabetic Foot Ulcers
Brief Title: Safety Study to Examine the Systemic Exposure of Granexin® Gel After Topical Application to Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xequel Bio, Inc. (Other)
Collaborators: Medical University of South Carolina (Other); Spartanburg Regional Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFU-PK-300
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Foot Ulcers
Keywords: Granexin; diabetic foot ulcers; pharmacokinetic study; FirstString Research
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Granexin® gel plus standard-of-care (Other): Granexin® gel will be applied topically to diabetic foot ulcer(s) on Day 0 (baseline), Day 3, and Day 7. In addition, standard-of-care treatment will be applied to the ulcer(s) at Screening, Day 0, Day 3, and Day 7.
  Interventions: Drug: Granexin® gel

INTERVENTIONS:
Drug: Granexin® gel — Granexin® gel will be dispensed directly from a 5 gram laminate tube and will be spread and smoothed directly over the wound surface in full contact with the wound bed to obtain an even, uniform layer on Day 0 (baseline), Day 3, and Day 7.

SUMMARY:
The purpose of this study is to determine the systemic exposure of Granexin® gel after topical application to human subjects' diabetic foot ulcers.

DETAILED DESCRIPTION:
The objective of this study is to ascertain the systemic exposure of the active ingredient in Granexin® gel (aCT1 peptide) after topical application to diabetic foot ulcers using pharmacokinetic analysis. It is planned that a total of 16 patients with diabetic foot ulcers will receive Granexin® gel treatment plus standard of care in this one arm study. The study includes a screening period (1 week) and a treatment period (1 week) which occur sequentially for a given patient. The baseline day, which demarcates the beginning of the treatment period, is the designated as Day 0. Screening procedures are initially conducted on Day -7.

A target foot ulcer is identified at screening and patient eligibility is confirmed at screening and then again at the beginning of the Day 0 (baseline) visit. A patient enrolled in the study may have multiple ulcers on the same or either foot; in this case, all ulcers will be treated with Granexin® gel, but only ulcer(s) meeting the following criteria will be designated as the target ulcer(s) and will determine eligibility: >4cm2 in post debridement of at least 4 weeks duration.

The treatment period for a given patient begins on Day 0 and ends one week later; the last scheduled day of the treatment period is designated as Day 7. During the treatment period, each patient is scheduled to receive topical treatment with study drug gel (3 applications total) administered by study staff at scheduled study site visits at each of the following time points: Day 0, Day 3, and Day 7. All patients, regardless of treatment assignment, also receive standard-of-care treatment at scheduled study visits during the treatment period.

Study drug pre-application blood samples will be collected from each patient at Day 0, Day 3, and Day 7. Study drug post-application blood samples will be collected at Day 0 and Day 7 at time points specified in the protocol. These blood samples will be shipped to a designated laboratory for pharmacokinetic analysis.

Safety will be assessed during the treatment period by monitoring adverse events, measuring vital signs at each visit, performing physical examinations, electrocardiograms (ECG), as well as pharmacokinetic (PK) blood analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Established diagnosis of diabetes mellitus (type I or II)
3. Glycosylated hemoglobin (HbA1c) value < 10.0% at the screening visit
4. Diagnosis of neuropathic foot ulcer(s)
5. Designated foot ulcer meets the following criteria at both the screening an baseline visits. If the patient has multiple ulcers, at least one ulcer must meet the following criteria at both the screening and baseline visits: a) Present for at least 4 weeks; b) Full-thickness cutaneous ulcer below the ankle surface; c) University of Texas grade A1; d) Area (after debridement) > 4 square cm; e) Viable, granulating wound (investigator discretion)
6. Ankle brachial index 0.7 to 1.3 at both the screening and baseline visits
7. Signed informed consent
8. Female patients of childbearing potential must have a negative pregnancy test at screening and must agree to use hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence throughout until 2 weeks after the last administration of study drug.

Exclusion Criteria:

1. Decrease in size of the designated target ulcer(s) by ≥ 30% during the 7-day screening period.
2. Impaired cognition determined by clinical investigator
3. Cannot tolerate the off-loading method or cannot comply with study-defined standard-of-care treatment.
4. Has an ulcer that meets any of the following criteria: a) Shows signs of severe clinical infection, defined as pus oozing from the ulcer site; b) Is positive for β-hemolytic streptococci upon culture; c) Has > 50% slough, significant necrotic tissue, bone, tendon, or capsule exposure; d) Is highly exuding (i.e., requires daily change of dressing)
5. Requires total contact cast
6. Ankle brachial pressure index <0.7 or > 1.3 or ankle systolic pressure <70 mmHg.
7. Has a systemic infection
8. Has any 1 of the following (only 1 of the 3 tests is required): a) On Doppler waveform analysis of the dorsalis pedis and posterior tibial arteries, a monophasic or biphasic flow (with loss of reverse flow) in either the artery of either foot; b) Toe: bracial index < 0.7 or > 1.3; c) Transcutaneous oxygen pressure < 40 mmHg
9. Presence of active systemic or local cancer or tumor of any king (exception: nonmelanoma skin cancer allowable at investigator discretion)
10. Congestive heart failure (New York Heart Association class II-IV) or coronary heart disease with ST segment elevation, myocardial infarction or coronary artery bypass graft, or percutaneous transluminal coronary angioplasty within the last 6 months.
11. Active osteomyelitis of the foot with the target ulcer(s)
12. Active connctive tissue disease
13. Acute Charcot's neuro-arthropathy as determined by clinical and/or radiographic examination.
14. Active treatment with systemic corticosteroids.
15. Previous or current radiation therapy to the distal lower extremity or likelihood to receive this therapy during study participation.
16. Pregnant or nursing.
17. Uncontrolled anemia (hemoglobin < 10 g/dL in females and < 12 g/dL in males).
18. Estimated glomerular filtration rate < 25 g/L.
19. Poor nutritional status, defined as an albumin < 25 g/L.
20. Significant peripheral edema as per investigator's discretion
21. Known inability or unavailability to complete required study visits during study participation.
22. A psychiatric condition (e.g., suicidal ideation) or chronic alcohol or drug abuse problem, determined from the patient's medical history, which in the opinion of the investigator, may pose a threat to patient compliance.
23. Use of a platelet-derived growth factor within 28 days before screening.
24. Use of any investigational drug or therapy within 28 days before screening.
25. Has any other factor which may, in the opinion of the investigator, compromise participation and/or follow-up in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Measurement of aCT1 peptide (Active Pharmaceutical Ingredient in Granexin) levels in blood | Day 0
Measurement of aCT1 peptide (Active Pharmaceutical Ingredient in Granexin) levels in blood | Day 3
Measurement of aCT1 peptide (Active Pharmaceutical Ingredient in Granexin) levels in blood | Day 7

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Aiyan Diabetes Center, Augusta, Georgia
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Salem VA Medical Center, Salem, Virginia